CLINICAL TRIAL: NCT05502484
Title: Potential Effectiveness of Integrative Dialectical Behavioural Therapy for Adults With Autism and the Role of Sensory Hyper- and Hyposensitivity and Interoceptive BOdy-Awareness in Self-Regulation Development
Brief Title: Development of Self-regulation by Dialectial Behavioural Therapy in Adults With Autism
Acronym: DASHBOARD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dimence mental health institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DASHBOARD
Record Dates: First submitted 2022-06-28; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-05

CONDITIONS: Autism Spectrum Disorder; Regulation, Self
Keywords: Autism Spectrum Disorder (ASD); dialectical behavioural therapy (DBT); self-regulation; emotion-dysregulation; body-awareness; interoception; sensory hypersensitivity; sensory hyposensitivity; non-suicidal self-injury (NSSI); suicidal ideation; suicidal behaviour; coping skills
MeSH Terms: conditions — Autism Spectrum Disorder; Self-Control; Self-Injurious Behavior; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Randomized multiple baseline design with staggered starts (randomized allocation to a baseline length of 4, 6, or 8 weeks) before starting the treatment (integrative Dialectical Behavioural Therapy).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 weeks baseline followed by Integrative DBT (Experimental): Integrative Dialectical Behavioural Therapy (DBT) consisting of 8 weeks outpatient pretreatment DBT, 40 weeks inpatient DBT, 24 weeks follow-up including 12 weeks after care DBT and 12 weeks no DBT.
  Interventions: Behavioral: Integrative Dialectical Behavioural Therapy (DBT)
- 6 weeks baseline followed by Integrative DBT (Experimental): Integrative Dialectical Behavioural Therapy (DBT) consisting of 8 weeks outpatient pretreatment DBT, 40 weeks inpatient DBT, 24 weeks follow-up including 12 weeks after care DBT and 12 weeks no DBT.
  Interventions: Behavioral: Integrative Dialectical Behavioural Therapy (DBT)
- 8 weeks baseline followed by Integrative DBT (Experimental): Integrative Dialectical Behavioural Therapy (DBT) consisting of 8 weeks outpatient pretreatment DBT, 40 weeks inpatient DBT, 24 weeks follow-up including 12 weeks after care DBT and 12 weeks no DBT.
  Interventions: Behavioral: Integrative Dialectical Behavioural Therapy (DBT)

INTERVENTIONS:
Behavioral: Integrative Dialectical Behavioural Therapy (DBT) — 8 weeks outpatient pre-treatment DBT followed by integrative, inpatient DBT of 40 weeks, using standard DBT, augmented with an experience-oriented, body-oriented skills training based on DBT-principles by trained DBT-therapists, and a follow-up phase of 12 weeks outpatient aftercare (maximal 8 sessions individual DBT and 4 booster sessions) and 12 weeks no DBT. The inpatient treatment takes place in a living environment that is based on the principles of DBT and takes into account several aspects of autism.

SUMMARY:
Individuals with autism spectrum disorder (ASD) are at risk to develop more pervasive emotion-dysregulation. In this study experiences of adults with ASD and severe emotion dysregulation with Integrative Dialectical Behaviour Therapy (DBT) and the mechanisms and processes that hinder and advance the pathway to recovery will be studied, in order to make the treatment more tailored and effective for this target group.

DETAILED DESCRIPTION:
Individuals with autism spectrum disorder (ASD) are at risk to develop more pervasive emotion-dysregulation and in conjunction with that they also show more maladaptive coping compared to non-autistic people. Sensory differences and impaired interoceptive body-awareness may influence emotion-dysregulation. Maladaptive coping is reflected by a variety of harmful behaviours, particularly strong social avoidance, rumination, obsessive-compulsive symptoms, disordered eating, substance abuse, agitation, non-suicidal-self-injury (NSSI), and suicidal ideation and behaviour. For a part of these individuals, treatment as usual does not have any effect at all, causing a vicious circle of isolation, demoralization, life-long psychiatric treatments, and crisis. DBT is an empirically supported psychotherapy to treat severe emotion-dysregulation. An effective inpatient treatment for adults with ASD and severe emotion-dysregulation is lacking, as well insight in the development of the process of self-regulation, particularly the role of sensory hyper- and hyposensitivity and interoceptive body-awareness. Therefore, an integrative, mostly inpatient treatment program based on DBT is developed and outcomes will be evaluated in the currently presented research. Standard DBT is used, adapted to adults with ASD, and augmented with a body-oriented DBT-skills training, because of their possible impairments of interoceptive body-awareness. Experiences of participants with the treatment program, the mechanisms and processes that hinder and advance the pathway to recovery will be studied, in order to make the treatment more tailored and effective for this target group.

The first aim is to quantify the effectiveness of integrative DBT in adults with ASD and difficult to treat severe emotion-dysregulation and maladaptive coping (primary outcome measure). The second aim is to determine the improvements over time in sensory hyper- and hyposensitivity, interoceptive body-awareness, cognitive and behavioural emotion-regulation, and well-being. Moreover, we will explore how (full and partial) responders, non-responders and deteriorators will differ with regard to autistic traits, PTSS-symptoms, sensory hyper- and hyposensitivity and interoceptive body-awareness. The third aim is to determine how qualitative findings regarding patients' experiences with integrative DBT enhance the deeper understanding of the quantitative clinical outcomes, in order to get insight in the process and sustainability of self-regulation, and to make the treatment more tailored and effective in the pathway to recovery.

A mixed-methods strategy consisting of three elements is executed:

1. A randomized, multiple-baseline single-case design with staggered baselines of 4, 6, or 8 weeks (randomized allocation) and daily measurements of emotion dysregulation.
2. A quasi-experimental design with 5 measurements with questionnaires at baseline (T0), start outpatient DBT pretreatment of 8 weeks (T1), start inpatient DBT of 40 weeks (T2), end inpatient DBT (T3), and end follow-up of 24 weeks (T4).
3. A qualitative study consisting of interviews with 30 participants.

ELIGIBILITY:
The inclusion criteria to enroll in the study are the same as the inclusion criteria for integrative DBT. Inclusion Criteria:

* Age ≥ 18 years old.
* A clinical diagnosis of ASD as diagnosed by a qualified health care professional (in Dutch: BIG registration).
* Non-responding to TAU (treatment as usual) for at least a year.
* IQ ≥ 85, based upon previous levels of education or previous IQ test, when available.
* Consent from the participant to record the DBT sessions on video or audio for supervision and assessing therapy integrity.
* Proficient in the Dutch language.
* Motivation to address problems through integrative DBT.
* Ability to work on treatment goals in collaboration with multiple therapists and counselors and to function in a group of maximal 8 adults with ASD.

Exclusion Criteria:

- Severe, current psychotic and manic symptoms, severe substance abuse disorder and eating disorder, requiring other specialized treatment first.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Maladaptive coping: using harmful behaviours | Change during inpatient treatment (phase C, 40 weeks)
  The diary card consists of four Likert scale questions related to standard categories in DBT, such as suicidality, NSSI, substance abuse, and in addition rumination. Scores for each of the constructs will be obtained on a range from 0 - 5: 0 = no urge until 5 = very much urge and a measure of performance of the maladaptive coping (no/yes).

SECONDARY OUTCOMES:
Non Suicidal Self Injury (NSSI) | Change: during baseline period (Phase A, randomized 4-6-8 weeks); during pre-treatment (Phase B, 8 weeks); during inpatient treatment (Phase C, 40 weeks); during follow-up (Phase D: 24 weeks)
  NSSI will be assessed by the Self-Injury Questionnaire-Treatment Related (SIQ-TR, Dutch version: Zelfverwondingsvragenlijst; Claes & Vandereycken, 2007). The SIQ-TR addresses five common forms of NSSI (scratching, bruising, cutting, burning and biting), the frequency, duration and pain experience of NSSI. There is an open question in which other self-injurious behaviour can be recorded, that is not standard mentioned (e.g., head banging).
Suicidal ideation | Change: during baseline period (Phase A, randomized 4-6-8 weeks); during pre-treatment (Phase B, 8 weeks); during inpatient treatment (Phase C, 40 weeks); during follow-up (Phase D: 24 weeks)
  Suicidal ideation will be assessed by the Suicidal Ideation Attributes Scale (SIDAS, Dutch version, Van Spijker et al., 2014). The SIDAS is a 5-item scale assessing frequency (item 1), controllability (item 2), closeness to attempt (item 3), distress (item 4), and interference with daily activities (item 5) on 10-point scales over the past month.
Interoceptive body-awareness | Change: during baseline period (Phase A, randomized 4-6-8 weeks); during pre-treatment (Phase B, 8 weeks); during inpatient treatment (Phase C, 40 weeks); during follow-up (Phase D: 24 weeks)
  Interoceptive body-awareness will be assessed by the Multidimensional Assessment of Interoceptive Awareness, Dutch version (MAIA-2, Mehling et al., 2018).
  The MAIA is a multidimensional self-report measure of interoceptive body-awareness consisting of 37 items and 8 scales: Noticing, not ignoring, not worrying, attention regulation, emotional awareness, self-regulation, listening, trusting.
Emotion-dysregulation | Change: during baseline period (Phase A, randomized 4-6-8 weeks); during pre-treatment (Phase B, 8 weeks); during inpatient treatment (Phase C, 40 weeks); during follow-up (Phase D: 24 weeks)
  Emotion-dysregulation will be assessed by the Difficulties in Emotion Regulation Scale (DERS, Gratz & Roemer, 2004; Dutch translation: Neumann & Koot, 2010).
  The DERS is an self-report measure consisting of 36 items, and designed to assess multiple aspects of emotion-dysregulation.
Cognitive emotion-regulation | Change: during baseline period (Phase A, randomized 4-6-8 weeks); during pre-treatment (Phase B, 8 weeks); during inpatient treatment (Phase C, 40 weeks); during follow-up (Phase D: 24 weeks)
  Cognitive emotion-regulation will be assessed by the Cognitive Emotion Regulation Questionnaire (CERQ, Garnefski et al., 2001; Garnefski, Kraaij & Spinhoven, 2002; Garnefski & Kraaij, 2006). The CERQ consists of 9 scales with 4 items each that can be answered on a 5-point Likert scale ranging from 0 (almost never) to 5 (almost always). For each subscale score the 4 items are added (range 4 to 20), indicating the extent to which a certain strategy is used. The CERQ subscales are: self-blame, other-blame, rumination, catastrophizing (more maladaptive strategies), and acceptance, positive refocusing, refocus on planning, positive reappraisal, putting into perspective (more adaptive strategies).
Behavioural emotion-regulation | Change: during baseline period (Phase A, randomized 4-6-8 weeks); during pre-treatment (Phase B, 8 weeks); during inpatient treatment (Phase C, 40 weeks); during follow-up (Phase D: 24 weeks)
  Behavioural emotion-regulation will be measured by the Behavioural Emotion Regulation Questionnaire (BERQ, Garnefski & Kraaij, 2019). The BERQ consists of 5 scales with 4 items each that can be answered on a 5-point Likert scale ranging from 0 (almost never) to 5 (almost always). For each subscale score the 4 items are added (range 4 to 20). The BERQ subscales are seeking distraction, actively approaching and seeking social support, and withdrawal and ignoring.
Sensory sensitivity | Change: during baseline period (Phase A, randomized 4-6-8 weeks); during pre-treatment (Phase B, 8 weeks); during inpatient treatment (Phase C, 40 weeks); during follow-up (Phase D: 24 weeks)
  Hyper- and hyposensitivity will be measured by the Dutch Glasgow Sensory Questionnaire (GSQ-NL) (Kuiper et al., 2019). It consists of 42 self-reported questions scored on a 5-point Likert scale ranging from 0 (never) to 4 (always). There are six items representing each modality (visual, auditory, gustatory, olfactory, tactile, vestibular and proprioception), half measuring hypersensitivity and half measuring hyposensitivity.
Well-being | Change: during baseline period (Phase A, randomized 4-6-8 weeks); during pre-treatment (Phase B, 8 weeks); during inpatient treatment (Phase C, 40 weeks); during follow-up (Phase D: 24 weeks)
  Well-being will be measured by the Mental Health Continuum - Short Form (MHC-SF, Dutch version). The MHC-SF comprises 14 items, which represent emotional well-being, psychological well-being, and social well-being. Respondents indicate the frequency of experienced feelings in the last month on a 6-point scale ranging from 0 (never) to 5 (every day).
Maladaptive coping: using harmful behaviours | Change: during baseline period (Phase A, randomized 4-6-8 weeks); during pre-treatment (Phase B, 8 weeks); during follow-up (Phase D: 24 weeks)
  The diary card consists of four Likert scale questions related to standard categories

CONTACTS AND LOCATIONS:
Overall Officials: Ella Lobregt-van Buuren, MSc, Principal Investigator — Dimence mental health institute; Nanda Lambregts-Rommelse, PhD, Study Chair — Radboud University Medical Center; Wouter Staal, PhD, Study Chair — Radboud University Medical Center; Lisette Verhoeven, PhD, Study Chair — Dr. Leo Kannerhuis; Peter Goossens, PhD, Study Chair — Dimence mental health institute
Locations (1):
- Dimence mental health institute, Deventer, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
see: https://dmp.radboudumc.nl/plans/93902
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After data are published, possibly in 2025.
Access Criteria: conditions for access to the data are described here:
  https://www.dimencegroep.nl/onderzoek/sites/default/files/documenten/richtlijn_databeheerplan_def_092018_0.pdf
URL: https://dmp.radboudumc.nl/plans/93902